CLINICAL TRIAL: NCT02501161
Title: A Clinical Trial Comparing Long Term Glycaemic Control of Insulin Degludec/Liraglutide (IDegLira) Versus Insulin Glargine Therapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: A 104 Week Clinical Trial Comparing Long Term Glycaemic Control of Insulin Degludec/Liraglutide (IDegLira) Versus Insulin Glargine Therapy in Subjects With Type 2 Diabetes Mellitus
Acronym: DUAL™ VIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4228; 2014-005639-15 (EudraCT Number); U1111-1165-3914 (Other: WHO)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide QD + OAD(s) (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- insulin glargine QD + OAD(s) (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Injected subcutaneously (under the skin) once daily for 104 weeks. Dose individually adjusted.
  Arms: Insulin degludec/liraglutide QD + OAD(s)
Drug: insulin glargine — Injected subcutaneously (under the skin) once daily for 104 weeks. Dose individually adjusted.
  Arms: insulin glargine QD + OAD(s)

SUMMARY:
This trial is conducted in Africa, Asia, Europe, North America and South America. The purpose is to compare long-term glycaemic control of insulin degludec/liraglutide (IDegLira) versus insulin glargine (IGlar) in insulin naïve subjects with type 2 diabetes mellitus inadequately controlled with oral anti diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Subjects diagnosed with type 2 diabetes mellitus
* HbA1c 7.0-11.0% (both inclusive) (53-97 mmol/mol) by central laboratory analysis
* Body mass index greater than or equal to 20 kg/m^2
* Insulin naïve subjects; however short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Stable daily dose(s) including any of the following antidiabetic drug(s)/regimens within 90 days prior to the day of screening: a) Biguanides (metformin greater than or equal to 1500 mg or maximum tolerated dose documented in the subject medical record), b) Other OAD(s) allowed: sulphonylurea, glinides, pioglitazone, and DPP4-inhibitors (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated dose as documented in subjects medical record)

Exclusion Criteria:

* Screening calcitonin greater than or equal to 50 ng/L
* Renal impairment estimated Glomerular Filtration Rate (eGFR) less than 60 ml/min/1.73 m2 as per CKD-EPI value to be defined as listed in the classification CKD-EPI using IDMS for serum creatinine measurement on the day of screening
* Impaired liver function, defined as ALAT or ASAT greater than or equal to 2.5 times upper limit of normal
* Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroid Carcinoma
* History of pancreatitis (acute or chronic)
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening
* Anticipated initiation or change in concomitant medications for more than 14 consecutive days or on a frequent basis known to affect weight or glucose metabolism (e.g. orlistat, thyroid hormones, corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry GCR, 1452, Study Director — Novo Nordisk A/S
Locations (123):
- United States (40):
  - Novo Nordisk Investigational Site, Muscle Shoals, Alabama
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Bermuda Dunes, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Lake Worth, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Mendoza
- Brazil (2):
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Porto Alegre
- Czechia (2):
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Dunaújváros
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Pécs
- India (11):
  - Novo Nordisk Investigational Site, Secunderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Rohtak, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
  - Novo Nordisk Investigational Site, Ẕerifin
- Italy (7):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Cittadella (PD)
  - Novo Nordisk Investigational Site, Negrar (VR)
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Verona
- Mexico (4):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Durango
- Norway (8):
  - Novo Nordisk Investigational Site, Bodø
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Hoenefoss
  - Novo Nordisk Investigational Site, Kløfta
  - Novo Nordisk Investigational Site, Lierskogen
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Tananger
- Poland (3):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Zabrze
- Russia (5):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Stavropol
- Slovakia (5):
  - Novo Nordisk Investigational Site, Prievidza
  - Novo Nordisk Investigational Site, Sabinov
  - Novo Nordisk Investigational Site, Trebišov
  - Novo Nordisk Investigational Site, Trenčín
  - Novo Nordisk Investigational Site, Trnava
- South Africa (8):
  - Novo Nordisk Investigational Site, Cosmo City, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, eMkhomazi, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Alberton
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Bursa
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Rize
  - Novo Nordisk Investigational Site, Samsun
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Angus
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Dudley
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Fife
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Rotherham
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, Wolverhampton

REFERENCES:
- [Result] Aroda VR, Gonzalez-Galvez G, Gron R, Halladin N, Haluzik M, Jermendy G, Kok A, Orsy P, Sabbah M, Sesti G, Silver R. Durability of insulin degludec plus liraglutide versus insulin glargine U100 as initial injectable therapy in type 2 diabetes (DUAL VIII): a multicentre, open-label, phase 3b, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Aug;7(8):596-605. doi: 10.1016/S2213-8587(19)30184-6. Epub 2019 Jun 9. PMID 31189519
- [Derived] Philis-Tsimikas A, Aroda VR, De Block C, Billings LK, Liebl A, Sivarathinasami R, D'Cruz JM, Lingvay I. Higher Derived Time in Range With IDegLira Versus Insulin Glargine U100 in People With Type 2 Diabetes. J Diabetes Sci Technol. 2024 May;18(3):653-659. doi: 10.1177/19322968221149041. Epub 2023 Jan 29. PMID 36710452
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 130 sites in Argentina (4),Czech Republic (4), Hungary (5), India (11), Israel (8), Italy (7), Mexico (4), Norway (7), Poland (3), Russian Federation (8), Slovakia (5), South Africa (10), Turkey (8), United Kingdom (9) and United States (37).
Pre-assignment Details: Participants were randomised in a 1:1 manner to receive either IDegLira or IGlar as an adjunct to oral anti-diabetic drugs (OADs). OADs allowed were: biguanides, sulphonylurea (SU), glinides, pioglitazone, and dipeptidyl peptidase-4 inhibitors (DPP4-inhibitors), though glinides and DPP4-inhibitors were not allowed as monotherapy or in combination.
Groups:
- Insulin Degludec/Liraglutide: Participants received subcutaneous (s.c.) injection of Insulin degludec/liraglutide (IDegLira) once daily up to 104 weeks. Participants received 10 dose steps (10 units IDeg/0.36 milligrams [mg] liraglutide) initially. The dose was then escalated twice weekly until the fasting plasma glucose (FPG) target between 4.0-5.0 millimoles per liter (mmol/L) (72-90 milligrams per deciliter [mg/dL]) was reached. The maximum dose was 50 dose steps (50 units IDeg/1.8 mg liraglutide).
- Insulin Glargine: Participants received s.c. injection of insulin glargine (IGlar) once daily up to 104 weeks. Participants received 10 units of IGlar initially. The dose was then escalated twice weekly until the FPG target between 4.0-5.0 mmol/L (72-90 mg/dL) was reached.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Started | 506 | 506
Exposed | 506 | 504
Completed | 484 | 481
Not Completed | 22 | 25
Not completed — Adverse Event | 2 | 6
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Insulin Degludec/Liraglutide: Participants received s.c. injection of IDegLira once daily up to 104 weeks. Participants received 10 dose steps (10 units IDeg/0.36 mg liraglutide) initially. The dose was then escalated twice weekly until the FPG target between 4.0-5.0 mmol/L (72-90 mg/dL) was reached. The maximum dose was 50 dose steps (50 units IDeg/1.8 mg liraglutide).
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine | Total
Number analyzed (Participants) | 506 | 506 | 1012
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (10.0) | 56.4 (10.1) | 56.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 231 | 457
  Male | 280 | 275 | 555
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 126 | 241
  Not Hispanic or Latino | 391 | 380 | 771
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 424 | 414 | 838
  Black or African American | 25 | 28 | 53
  Asian | 54 | 61 | 115
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomisation to Inadequate Glycaemic Control and Need for Treatment Intensification
Description: Inadequate glycaemic control and need for treatment intensification was defined as a glycosylated haemoglobin (HbA1c) of 7.0% or greater at 2 consecutive visits from week 26, including week 26 if HbA1c was greater than or equal to 7% at week 12. Time from randomisation to inadequate glycaemic control and need for treatment intensification was analysed using a stratified log-rank test where treatment, baseline HbA1c group and previous OAD treatment were included as strata in the model. The variable "baseline HbA1c group" was a dichotomised baseline HbA1c variable with 2 categories: HbA1c < 8.5% or HbA1c ≥ 8.5% and the variable "previous OAD treatment" was a categorical variable with 2 categories: SU ± OAD(s) (SU users) or OAD(s) (Non-SU users). 25%, median (50%) and 75% percentiles for the cumulative distribution function were obtained from the Kaplan-Meier survival function.
Time Frame: Weeks 0-104 + 7 days follow-up-1 + 30 days follow-up-2
Population: FAS included all randomised participants. Number analyzed=participants in the specified category.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Weeks
  Baseline HbA1c <8.5% + Non-SU users: number analyzed (Participants) | 112 | 105
  Baseline HbA1c <8.5% + Non-SU users | NA [104.0 to NA] — The estimated median and 75 percentile data were not available as the proportions were not reached within study period. | 104.3 [38.1 to NA] — The 75 percentile data was not available as the proportions was not reached within study period.
  Baseline HbA1c <8.5% + SU users: number analyzed (Participants) | 185 | 135
  Baseline HbA1c <8.5% + SU users | 106.7 [89.9 to NA] — The 75 percentile data was not available as the proportions was not reached within study period. | 90.3 [26.4 to 105.1]
  Baseline HbA1c >=8.5% + Non-SU users: number analyzed (Participants) | 74 | 67
  Baseline HbA1c >=8.5% + Non-SU users | NA [39.7 to NA] — The estimated median and 75 percentile data were not available as the proportions were not reached within study period. | 64.6 [26.1 to 105.1]
  Baseline HbA1c >=8.5% + SU users: number analyzed (Participants) | 135 | 199
  Baseline HbA1c >=8.5% + SU users | 104.0 [26.4 to NA] — The 75 percentile data was not available as the proportions was not reached within study period. | 26.6 [26.1 to 91.1]
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Glargine; Test for no treatment difference was based on using a stratified log-rank test where treatment, baseline HbA1c group and pre-trial OAD treatment group were included as strata in the model; Test type: Other; p < .0001, Stratified log-rank test

2. Secondary Outcome: Time From Randomisation to HbA1c >6.5% at 2 Consecutive Visits
Description: Time to HbA1c > 6.5% at 2 consecutive visits is defined as time from randomization to HbA1c > 6.5% at 2 consecutive planned scheduled visits from week 26 (including week 26 if HbA1c was > 6.5% at week 12). Time from randomisation to HbA1c >6.5% at 2 consecutive visits was analysed using a stratified log-rank test where treatment, baseline HbA1c group and previous OAD treatment were included as strata in the model. The variable "baseline HbA1c group" was a dichotomised baseline HbA1c variable with 2 categories: HbA1c < 8.5% or HbA1c ≥ 8.5% and the variable "previous OAD treatment" was a categorical variable with 2 categories: SU ± OAD(s) (SU users) or OAD(s) (Non-SU users). 25%, median (50%) and 75% percentiles for the cumulative distribution function were obtained from the Kaplan-Meier survival function.
Time Frame: Weeks 0-104 + 7 days follow-up-1 + 30 days follow-up-2
Population: FAS included all randomised participants. Number analyzed=participants with event.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Weeks
  Baseline HbA1c <8.5% + Non-SU users: number analyzed (Participants) | 112 | 105
  Baseline HbA1c <8.5% + Non-SU users | NA [52.1 to NA] — The estimated median and 75 percentile data were not available as the proportions were not reached within study period. | 64.1 [26.1 to 104.3]
  Baseline HbA1c <8.5% + SU users: number analyzed (Participants) | 185 | 135
  Baseline HbA1c <8.5% + SU users | 90.1 [27.0 to NA] — The 75 percentile data was not available as the proportion was not reached within study period. | 26.6 [26.1 to 89.9]
  Baseline HbA1c >=8.5% + Non-SU users: number analyzed (Participants) | 74 | 67
  Baseline HbA1c >=8.5% + Non-SU users | 64.1 [26.1 to NA] — The 75 percentile data was not available as the proportion was not reached within study period. | 26.6 [26.1 to 90.1]
  Baseline HbA1c >=8.5% + SU users: number analyzed (Participants) | 135 | 199
  Baseline HbA1c >=8.5% + SU users | 52.1 [26.1 to 104.1] | 26.1 [26.1 to 38.1]
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Glargine; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, Stratified log-rank test

3. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of HbA1c | -1.99 (1.14) | -1.69 (1.10)

4. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Kilogram (kg)
  Week 26: number analyzed (Participants) | 481 | 466
  Week 26 | 0.5 (3.3) | 2.2 (3.6)
  Week 104: number analyzed (Participants) | 335 | 190
  Week 104 | 1.2 (4.9) | 3.0 (4.9)

5. Secondary Outcome: Insulin Dose
Description: Insulin dose after 26 and 104 weeks of treatment is presented.
Time Frame: Week 26, week 104
Population: Safety analysis set (SAS) included all participants receiving at least 1 dose of the investigational product (IDegLira) or comparator (IGlar). 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Units
  Week 26: number analyzed (Participants) | 476 | 449
  Week 26 | 34.6 (13.4) | 48.6 (28.2)
  Week 104: number analyzed (Participants) | 329 | 186
  Week 104 | 36.1 (12.9) | 50.6 (31.5)

6. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c <7.0%
Description: Percentage of participants who achieved (yes/no) HbA1c <7.0% at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 78.7 | 55.7
  Week 26: No | 21.3 | 44.3
  Week 104: Yes | 55.5 | 28.5
  Week 104: No | 44.5 | 71.5

7. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c <7.0% Without Weight Gain
Description: Percentage of participants who achieved (yes/no) HbA1c <7.0% without weight gain at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 38.5 | 15.4
  Week 26: No | 61.5 | 84.6
  Week 104: Yes | 20.9 | 6.3
  Week 104: No | 79.1 | 93.7

8. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c <7.0% Without Treatment-emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemia was defined as an episode that was severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Percentage of participants who achieved (yes/no) HbA1c <7.0% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 71.3 | 44.9
  Week 26: No | 28.7 | 55.1
  Week 104: Yes | 51.8 | 25.5
  Week 104: No | 48.2 | 74.5

9. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c < 7.0% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes and Without Weight Gain
Description: Severe or BG confirmed symptomatic hypoglycaemia was defined as an episode that was severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Percentage of participants who achieved (yes/no) HbA1c <7.0% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes and without weight gain at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 35.2 | 13.6
  Week 26: No | 64.8 | 86.4
  Week 104: Yes | 20.0 | 6.1
  Week 104: No | 80.0 | 93.9

10. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c ≤6.5%
Description: Percentage of participants who achieved (yes/no) HbA1c ≤6.5% at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 63.6 | 35.4
  Week 26: No | 36.4 | 64.6
  Week 104: Yes | 43.3 | 21.7
  Week 104: No | 56.7 | 78.3

11. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c ≤6.5% Without Weight Gain
Description: Percentage of participants who achieved (yes/no) HbA1c ≤6.5% without weight gain at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 33.2 | 9.9
  Week 26: No | 66.8 | 90.1
  Week 104: Yes | 17.6 | 5.7
  Week 104: No | 82.4 | 94.3

12. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c ≤6.5% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Percentage of participants who achieved (yes/no) HbA1c ≤6.5% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 57.9 | 27.9
  Week 26: No | 42.1 | 72.1
  Week 104: Yes | 40.1 | 19.2
  Week 104: No | 59.9 | 80.8

13. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c ≤6.5% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes and Without Weight Gain
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Percentage of participants who achieved (yes/no) HbA1c ≤6.5% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes and without weight gain at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Percentage of participants
  Week 26: Yes | 30.2 | 8.7
  Week 26: No | 69.8 | 91.3
  Week 104: Yes | 16.6 | 5.5
  Week 104: No | 83.4 | 94.5

14. Secondary Outcome: Change in FPG
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
mmol/L
  Week 26: number analyzed (Participants) | 475 | 461
  Week 26 | -3.97 (3.06) | -3.79 (3.18)
  Week 104: number analyzed (Participants) | 328 | 185
  Week 104 | -3.93 (2.96) | -3.73 (2.75)

15. Secondary Outcome: SMPG-9-point Profile (Individual Points in the Profile)
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. Self-measured plasma glucose (SMPG)-9-point profile (individual points in the profile) at week 26 and week 104 is presented.
Time Frame: Week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
mmol/L
  Week 26: Before breakfast: number analyzed (Participants) | 437 | 413
  Week 26: Before breakfast | 5.59 (1.57) | 5.58 (1.58)
  Week 26: 90 minutes after breakfast: number analyzed (Participants) | 425 | 409
  Week 26: 90 minutes after breakfast | 8.34 (2.62) | 8.76 (2.68)
  Week 26: Before lunch: number analyzed (Participants) | 435 | 407
  Week 26: Before lunch | 6.03 (2.00) | 6.43 (2.24)
  Week 26: 90 minutes after lunch: number analyzed (Participants) | 433 | 407
  Week 26: 90 minutes after lunch | 8.02 (2.32) | 8.79 (2.64)
  Week 26: Before dinner: number analyzed (Participants) | 434 | 408
  Week 26: Before dinner | 6.67 (2.26) | 6.91 (2.35)
  Week 26: 90 minutes after dinner: number analyzed (Participants) | 428 | 406
  Week 26: 90 minutes after dinner | 8.31 (2.47) | 9.10 (2.70)
  Week 26: Bedtime: number analyzed (Participants) | 423 | 398
  Week 26: Bedtime | 7.48 (2.42) | 8.13 (2.68)
  Week 26: At 4:00 a.m.: number analyzed (Participants) | 419 | 398
  Week 26: At 4:00 a.m. | 5.72 (1.55) | 5.91 (1.99)
  Week 26: Before breakfast the following day: number analyzed (Participants) | 433 | 403
  Week 26: Before breakfast the following day | 5.53 (1.37) | 5.56 (1.56)
  Week 104: Before breakfast: number analyzed (Participants) | 296 | 171
  Week 104: Before breakfast | 5.58 (1.38) | 5.57 (1.27)
  Week 104: 90 minutes after breakfast: number analyzed (Participants) | 287 | 166
  Week 104: 90 minutes after breakfast | 7.99 (2.50) | 8.64 (2.59)
  Week 104: Before lunch: number analyzed (Participants) | 290 | 167
  Week 104: Before lunch | 6.06 (1.91) | 6.37 (2.02)
  Week 104: 90 minutes after lunch: number analyzed (Participants) | 290 | 167
  Week 104: 90 minutes after lunch | 7.80 (2.16) | 8.87 (2.45)
  Week 104: Before dinner: number analyzed (Participants) | 292 | 168
  Week 104: Before dinner | 6.58 (1.97) | 7.02 (2.45)
  Week 104: 90 minutes after dinner: number analyzed (Participants) | 290 | 167
  Week 104: 90 minutes after dinner | 8.20 (2.20) | 9.10 (2.61)
  Week 104: Bedtime: number analyzed (Participants) | 286 | 164
  Week 104: Bedtime | 7.47 (2.17) | 7.90 (2.41)
  Week 104: At 4:00 a.m.: number analyzed (Participants) | 284 | 163
  Week 104: At 4:00 a.m. | 5.67 (1.35) | 5.96 (1.73)
  Week 104: Before breakfast the following day: number analyzed (Participants) | 292 | 169
  Week 104: Before breakfast the following day | 5.44 (1.23) | 5.47 (1.35)

16. Secondary Outcome: Change in SMPG-mean 9-point Profile
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. Change in SMPG-mean 9-point profile from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
mmol/L
  Week 26: number analyzed (Participants) | 422 | 389
  Week 26 | -3.34 (2.46) | -3.32 (2.62)
  Week 104: number analyzed (Participants) | 285 | 161
  Week 104 | -3.27 (2.36) | -2.76 (2.41)

17. Secondary Outcome: Change in SMPG-mean Postprandial Increment Over All Meals
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. Change in SMPG-mean postprandial increment over all meals from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
mmol/L
  Week 26: number analyzed (Participants) | 428 | 405
  Week 26 | -0.28 (2.13) | 0.20 (2.17)
  Week 104: number analyzed (Participants) | 286 | 164
  Week 104 | -0.47 (1.99) | 0.12 (2.17)

18. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic)
Description: Change in blood pressure (systolic and diastolic) from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Millimeters of mercury (mmHg)
  Week 26: Systolic blood pressure: number analyzed (Participants) | 482 | 466
  Week 26: Systolic blood pressure | -1.2 (14.0) | 0.5 (13.1)
  Week 26: Diastolic blood pressure: number analyzed (Participants) | 482 | 466
  Week 26: Diastolic blood pressure | 0.1 (8.8) | -0.3 (8.4)
  Week 104: Systolic blood pressure: number analyzed (Participants) | 335 | 190
  Week 104: Systolic blood pressure | 0.5 (14.3) | 0.9 (13.6)
  Week 104: Diastolic blood pressure: number analyzed (Participants) | 335 | 190
  Week 104: Diastolic blood pressure | -0.1 (8.8) | -0.2 (8.6)

19. Secondary Outcome: Change in Fasting C-peptide
Description: Change in fasting C-peptide (measured in nanomoles per liter [nmol/L]) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-peptide
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of C-peptide
  Week 26: number analyzed (Participants) | 474 | 458
  Week 26 | 0.63 (60.79) | 0.57 (62.44)
  Week 104: number analyzed (Participants) | 333 | 184
  Week 104 | 0.58 (64.21) | 0.54 (70.45)

20. Secondary Outcome: Change in Fasting Human Insulin
Description: Change in fasting human insulin (measured in picomoles per liter [pmol/L]) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of insulin
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of insulin
  Week 26: number analyzed (Participants) | 478 | 456
  Week 26 | 0.67 (90.68) | 0.68 (89.19)
  Week 104: number analyzed (Participants) | 330 | 186
  Week 104 | 0.60 (91.84) | 0.62 (92.55)

21. Secondary Outcome: Change in Fasting Total Cholesterol
Description: Change in fasting total cholesterol (measured in mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 470 | 455
  Week 26 | 0.99 (17.38) | 0.99 (17.68)
  Week 104: number analyzed (Participants) | 319 | 181
  Week 104 | 0.97 (19.11) | 0.97 (20.40)

22. Secondary Outcome: Change in Fasting LDL-cholesterol
Description: Change in fasting low density lipoprotein (LDL)-cholesterol (measured in mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL-cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of LDL-cholesterol
  Week 26: number analyzed (Participants) | 467 | 452
  Week 26 | 1.05 (35.97) | 1.02 (30.10)
  Week 104: number analyzed (Participants) | 318 | 178
  Week 104 | 0.96 (38.83) | 0.98 (34.40)

23. Secondary Outcome: Change in Fasting HDL-cholesterol
Description: Change in fasting high density lipoprotein (HDL)- cholesterol (measured in mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL-cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of HDL-cholesterol
  Week 26: number analyzed (Participants) | 467 | 454
  Week 26 | 1.03 (16.61) | 1.02 (15.57)
  Week 104: number analyzed (Participants) | 319 | 180
  Week 104 | 1.02 (16.93) | 1.03 (17.36)

24. Secondary Outcome: Change in Fasting VLDL-cholesterol
Description: Change in fasting very low density lipoprotein (VLDL)-cholesterol (measured in mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL-cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of VLDL-cholesterol
  Week 26: number analyzed (Participants) | 468 | 453
  Week 26 | 0.85 (40.78) | 0.85 (42.01)
  Week 104: number analyzed (Participants) | 318 | 179
  Week 104 | 0.90 (40.90) | 0.88 (35.98)

25. Secondary Outcome: Change in Fasting Triglycerides
Description: Change in fasting triglycerides (measured as mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 469 | 455
  Week 26 | 0.84 (43.82) | 0.85 (45.75)
  Week 104: number analyzed (Participants) | 319 | 181
  Week 104 | 0.89 (42.20) | 0.89 (40.08)

26. Secondary Outcome: Change in Fasting Free Fatty Acids
Description: Change in fasting free fatty acids (measured as mmol/L) from baseline (week 0) to week 26 and week 104 is presented as ratio to baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Ratio of free fatty acids
  Week 26: number analyzed (Participants) | 474 | 460
  Week 26 | 0.68 (59.69) | 0.75 (60.25)
  Week 104: number analyzed (Participants) | 332 | 186
  Week 104 | 0.70 (57.71) | 0.78 (59.48)

27. Secondary Outcome: Number of Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During 26 Weeks of Treatment
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during 26 weeks of treatment is presented.
Time Frame: Weeks 0-26
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 143 | 261

28. Secondary Outcome: Number of Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During 104 Weeks of Treatment
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during 104 weeks of treatment is presented.
Time Frame: Weeks 0-104
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 319 | 642

29. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes During 26 Weeks of Treatment
Description: Hypoglycaemic episodes (SMPG value ≤3.9 mmol/L (70 mg/dL)) were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent hypoglycaemic episodes according to ADA during 26 weeks of treatment is presented.
Time Frame: Weeks 0-26
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 3190 | 3806

30. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes During 104 Weeks of Treatment
Description: Hypoglycaemic episodes (SMPG value ≤3.9 mmol/L (70 mg/dL)) were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment emergent hypoglycaemic episodes according to ADA during 104 weeks of treatment is presented.
Time Frame: Weeks 0-104
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 8934 | 10658

31. Secondary Outcome: Number of Treatment-emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During 26 Weeks of Treatment
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Nocturnal hypoglycaemic episodes were episodes occurring between 00:01 and 05.59 both inclusive. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes during 26 weeks of treatment is presented.
Time Frame: Weeks 0-26
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 27 | 60

32. Secondary Outcome: Number of Treatment-emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During 104 Weeks of Treatment
Description: Severe or BG confirmed symptomatic hypoglycaemia is defined as an episode that is severe according to the ADA classification or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Nocturnal hypoglycaemic episodes were episodes occurring between 00:01 and 05.59 both inclusive. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes during 104 weeks of treatment is presented.
Time Frame: Weeks 0-104
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Episodes | 61 | 164

33. Secondary Outcome: Number of TEAEs During 26 Weeks of Treatment
Description: An adverse event is any untoward medical occurrence in a participant administered a product, and which does not necessarily have a causal relationship with this treatment. A treatment emergent adverse event (TEAE) was defined as an adverse event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product. If the event had onset date before the first day of exposure on trial product and increased in severity during the treatment period and until 7 days after the last drug date, then this event was also considered as a TEAE. Number of TEAEs during 26 weeks of treatment is presented.
Time Frame: Weeks 0-26
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Adverse events
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Adverse events | 718 | 624

34. Secondary Outcome: Number of TEAEs During 104 Weeks of Treatment
Description: An adverse event is any untoward medical occurrence in a participant administered a product, and which does not necessarily have a causal relationship with this treatment. A TEAE was defined as an adverse event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product. If the event had onset date before the first day of exposure on trial product and increased in severity during the treatment period and until 7 days after the last drug date, then this event was also considered as a TEAE. Number of TEAEs during 104 weeks of treatment is presented.
Time Frame: Week 0 to week 104
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator.
Measure: Number; unit: Adverse events
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Adverse events | 1788 | 1368

35. Secondary Outcome: Eye Examination Category
Description: Fundus photography or a dilated fundoscopy was performed at baseline (within 12 weeks prior to week 0) and week 104. The investigator interpreted each eye's (left and right) results and categorised them as: normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). Number of participants in each category at baseline and week 104 were presented.
Time Frame: Baseline (within 12 weeks prior to week 0), week 104
Population: SAS included all participants receiving at least 1 dose of the investigational product or comparator. 'Number analyzed'=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Participants
  Left eye: Normal (baseline) | 345 | 341
  Left eye: Abnormal NCS (baseline) | 151 | 155
  Left eye: Abnormal CS (baseline) | 10 | 8
  Left eye: Normal (week 104): number analyzed (Participants) | 318 | 185
  Left eye: Normal (week 104) | 204 | 129
  Left eye: Abnormal NCS (week 104): number analyzed (Participants) | 318 | 185
  Left eye: Abnormal NCS (week 104) | 97 | 50
  Left eye: Abnormal CS (week 104): number analyzed (Participants) | 318 | 185
  Left eye: Abnormal CS (week 104) | 17 | 6
  Right eye: Normal (baseline) | 344 | 355
  Right eye: Abnormal NCS (baseline) | 151 | 143
  Right eye: Abnormal CS (baseline) | 11 | 6
  Right eye: Normal (week 104): number analyzed (Participants) | 318 | 185
  Right eye: Normal (week 104) | 200 | 132
  Right eye: Abnormal NCS (week 104): number analyzed (Participants) | 318 | 185
  Right eye: Abnormal NCS (week 104) | 99 | 48
  Right eye: Abnormal CS (week 104): number analyzed (Participants) | 318 | 185
  Right eye: Abnormal CS (week 104) | 19 | 5

36. Secondary Outcome: ECG Evaluation
Description: The electrocardiogram (ECG) was assessed at baseline (within 2 weeks prior to week 0) and week 104. The investigator interpreted the results and categorised them as: normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline and week 104 are presented.
Time Frame: Baseline (within 2 weeks prior to week 0), week 104
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Participants
  Normal (Baseline) | 335 | 335
  Abnormal NCS (Baseline) | 162 | 165
  Abnormal CS (Baseline) | 9 | 4
  Normal (week 104): number analyzed (Participants) | 331 | 189
  Normal (week 104) | 227 | 122
  Abnormal NCS (week 104): number analyzed (Participants) | 331 | 189
  Abnormal NCS (week 104) | 97 | 65
  Abnormal CS (week 104): number analyzed (Participants) | 331 | 189
  Abnormal CS (week 104) | 7 | 2

37. Secondary Outcome: Change in Urine Albumin/Creatinine Ratio
Description: Change in urine albumin/creatinine ratio from baseline (week 0) to week 104 is presented.
Time Frame: Week 0, week 104
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Milligrams per millimole (mg/mmol)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Milligrams per millimole (mg/mmol) | -1.09 (7.43) | -0.74 (15.58)

38. Secondary Outcome: Change in Pulse Rate
Description: Change in pulse rate from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: SAS included all participants who received at least 1 dose of the investigational product or comparator. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Beats per minute
  Week 26: number analyzed (Participants) | 482 | 466
  Week 26 | 2.0 (8.8) | -0.4 (8.7)
  Week 104: number analyzed (Participants) | 335 | 189
  Week 104 | 1.7 (9.3) | -0.5 (9.7)

39. Secondary Outcome: Change in Biochemistry Parameter- Creatinine, Total Bilirubin
Description: Change in biochemistry parameter- creatinine, total bilirubin from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Micromoles per liter (umol/L)
  Week 26: creatinine: number analyzed (Participants) | 476 | 462
  Week 26: creatinine | -0.50 (10.08) | 0.25 (8.78)
  Week 104: creatinine: number analyzed (Participants) | 325 | 184
  Week 104: creatinine | 0.75 (10.85) | 2.20 (11.86)
  Week 26: total bilirubin: number analyzed (Participants) | 476 | 462
  Week 26: total bilirubin | -0.30 (3.35) | -0.32 (2.80)
  Week 104: total bilirubin: number analyzed (Participants) | 324 | 182
  Week 104: total bilirubin | -0.33 (3.42) | -0.59 (3.01)

40. Secondary Outcome: Change in Biochemistry Parameter- Albumin
Description: Change in biochemistry parameter- albumin from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Grams per deciliter (g/dL)
  Week 26: number analyzed (Participants) | 477 | 462
  Week 26 | -0.03 (0.24) | -0.03 (0.21)
  Week 104: number analyzed (Participants) | 324 | 184
  Week 104 | 0.01 (0.24) | 0.03 (0.27)

41. Secondary Outcome: Change in Biochemistry Parameters- ALP, ALT, AST, Lipase and Amylase
Description: Change in biochemistry parameters- alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lipase and amylase from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Units per liter (U/L)
  Week 26: ALP: number analyzed (Participants) | 476 | 462
  Week 26: ALP | -4.16 (14.16) | -4.33 (12.84)
  Week 104: ALP: number analyzed (Participants) | 324 | 183
  Week 104: ALP | -1.35 (15.71) | -1.34 (14.22)
  Week 26: ALT: number analyzed (Participants) | 476 | 462
  Week 26: ALT | -5.45 (18.50) | -3.33 (13.24)
  Week 104: ALT: number analyzed (Participants) | 323 | 184
  Week 104: ALT | -5.39 (14.16) | -3.45 (14.46)
  Week 26: AST: number analyzed (Participants) | 476 | 462
  Week 26: AST | -1.62 (9.78) | -0.39 (9.51)
  Week 104: AST: number analyzed (Participants) | 323 | 182
  Week 104: AST | -1.84 (9.86) | -0.67 (10.78)
  Week 26: lipase: number analyzed (Participants) | 476 | 462
  Week 26: lipase | 9.26 (42.92) | -7.97 (34.28)
  Week 104: lipase: number analyzed (Participants) | 325 | 184
  Week 104: lipase | 5.41 (48.35) | -13.33 (42.27)
  Week 26: amylase: number analyzed (Participants) | 477 | 462
  Week 26: amylase | 9.72 (23.28) | 2.79 (20.92)
  Week 104: amylase: number analyzed (Participants) | 325 | 184
  Week 104: amylase | 7.23 (25.42) | -0.13 (25.94)

42. Secondary Outcome: Change in Biochemistry Parameter- Sodium, Potassium and Calcium
Description: Change in sodium, potassium and calcium from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
mmol/L
  Week 26: sodium: number analyzed (Participants) | 477 | 462
  Week 26: sodium | 0.89 (2.74) | 1.03 (2.61)
  Week 104: sodium: number analyzed (Participants) | 325 | 184
  Week 104: sodium | 1.22 (2.54) | 1.47 (2.39)
  Week 26: potassium: number analyzed (Participants) | 477 | 461
  Week 26: potassium | -0.05 (0.40) | -0.08 (0.42)
  Week 104: potassium: number analyzed (Participants) | 324 | 184
  Week 104: potassium | -0.06 (0.42) | -0.07 (0.43)
  Week 26: calcium: number analyzed (Participants) | 475 | 462
  Week 26: calcium | -0.01 (0.11) | -0.00 (0.11)
  Week 104: calcium: number analyzed (Participants) | 323 | 184
  Week 104: calcium | -0.07 (0.10) | -0.06 (0.11)

43. Secondary Outcome: Change in Haematological Parameter- Haemoglobin
Description: Change in haemoglobin from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
g/dL
  Week 26: number analyzed (Participants) | 480 | 463
  Week 26 | 0.08 (0.72) | 0.08 (0.74)
  Week 104: number analyzed (Participants) | 331 | 185
  Week 104 | -0.00 (0.89) | -0.03 (0.92)

44. Secondary Outcome: Change in Haematological Parameter- Haematocrit
Description: Change in haematocrit from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of red blood cells
  Week 26: number analyzed (Participants) | 478 | 462
  Week 26 | -0.33 (2.45) | -0.36 (2.43)
  Week 104: number analyzed (Participants) | 329 | 184
  Week 104 | -0.71 (2.83) | -0.95 (3.02)

45. Secondary Outcome: Change in Haematological Parameter- Erythrocytes
Description: Change in erythrocytes from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
10^12 cells/L
  Week 26: number analyzed (Participants) | 480 | 464
  Week 26 | -0.02 (0.28) | -0.03 (0.27)
  Week 104: number analyzed (Participants) | 331 | 185
  Week 104 | -0.12 (0.30) | -0.11 (0.32)

46. Secondary Outcome: Change in Haematological Parameter- Thrombocytes and Leukocytes
Description: Change in thrombocytes and leukocytes from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
10^9 cells/L
  Week 26: Thrombocytes: number analyzed (Participants) | 476 | 463
  Week 26: Thrombocytes | 8.77 (35.82) | 7.05 (41.71)
  Week 104: Thrombocytes: number analyzed (Participants) | 326 | 184
  Week 104: Thrombocytes | 16.87 (39.27) | 18.73 (53.76)
  Week 26: Leukocytes: number analyzed (Participants) | 480 | 464
  Week 26: Leukocytes | 0.49 (1.45) | 0.39 (1.43)
  Week 104: Leukocytes: number analyzed (Participants) | 329 | 185
  Week 104: Leukocytes | 0.07 (1.50) | 0.32 (1.55)

47. Secondary Outcome: Change in Haematological Parameter- Eosinophils
Description: Change in eosinophils from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of eosinophils
  Week 26: number analyzed (Participants) | 478 | 464
  Week 26 | 0.10 (1.88) | 0.06 (2.09)
  Week 104: number analyzed (Participants) | 326 | 183
  Week 104 | 0.32 (2.08) | 0.43 (1.56)

48. Secondary Outcome: Change in Haematological Parameter- Neutrophils
Description: Change in neutrophils from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of neutrophils
  Week 26: number analyzed (Participants) | 478 | 464
  Week 26 | 1.86 (7.20) | 0.78 (7.68)
  Week 104: number analyzed (Participants) | 326 | 183
  Week 104 | 1.25 (7.94) | 1.21 (8.02)

49. Secondary Outcome: Change in Haematological Parameter- Basophils
Description: Change in basophils from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of basophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of basophils
  Week 26: number analyzed (Participants) | 478 | 464
  Week 26 | 0.00 (0.28) | -0.00 (0.29)
  Week 104: number analyzed (Participants) | 326 | 183
  Week 104 | 0.20 (0.38) | 0.16 (0.35)

50. Secondary Outcome: Change in Haematological Parameter- Monocytes
Description: Change in monocytes from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of monocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of monocytes
  Week 26: number analyzed (Participants) | 478 | 464
  Week 26 | -0.10 (2.04) | 0.01 (1.91)
  Week 104: number analyzed (Participants) | 326 | 183
  Week 104 | 0.49 (2.02) | 0.59 (1.88)

51. Secondary Outcome: Change in Haematological Parameter- Lymphocytes
Description: Change in lymphocytes from baseline (week 0) to week 26 and week 104 is presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Percentage of lymphocytes
  Week 26: number analyzed (Participants) | 478 | 464
  Week 26 | -1.87 (6.29) | -0.84 (6.73)
  Week 104: number analyzed (Participants) | 326 | 183
  Week 104 | -2.25 (6.76) | -2.38 (7.29)

52. Secondary Outcome: Change in Calcitonin
Description: The number of participants who reported low, normal and high levels of calcitonin in relation to reference ranges at baseline (week 0), week 26 and week 104 are presented.
Time Frame: Week 0, week 26, week 104
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 504
Participants
  Week 0: Low | 0 | 0
  Week 0: Normal | 481 | 472
  Week 0: High | 25 | 32
  Week 26: Low: number analyzed (Participants) | 477 | 461
  Week 26: Low | 0 | 0
  Week 26: Normal: number analyzed (Participants) | 477 | 461
  Week 26: Normal | 437 | 431
  Week 26: High: number analyzed (Participants) | 477 | 461
  Week 26: High | 40 | 30
  Week 104: Low: number analyzed (Participants) | 332 | 186
  Week 104: Low | 0 | 0
  Week 104: Normal: number analyzed (Participants) | 332 | 186
  Week 104: Normal | 301 | 169
  Week 104: High: number analyzed (Participants) | 332 | 186
  Week 104: High | 31 | 17

53. Secondary Outcome: Change in Short Form Health Survey Version 2.0 (SF-36v2™, Acute Version) Health Survey: Scores From the 8 Domains and Summaries of the Physical Component Score (PCS) and the Mental Component Score (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in the sub-domain scores and component summary (PCS and MCS) scores are presented. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Score on a scale
  Week 26: Physical functioning: number analyzed (Participants) | 482 | 465
  Week 26: Physical functioning | 1.2 (6.8) | 1.1 (7.0)
  Week 104: Physical functioning: number analyzed (Participants) | 335 | 190
  Week 104: Physical functioning | 0.7 (7.5) | 0.6 (7.9)
  Week 26: Role-physical: number analyzed (Participants) | 482 | 465
  Week 26: Role-physical | 1.4 (7.7) | 0.5 (7.4)
  Week 104: Role-physical: number analyzed (Participants) | 335 | 190
  Week 104: Role-physical | 1.4 (8.7) | 0.7 (7.5)
  Week 26: Bodily pain: number analyzed (Participants) | 482 | 465
  Week 26: Bodily pain | 1.5 (9.7) | 0.4 (10.0)
  Week 104: Bodily pain: number analyzed (Participants) | 335 | 190
  Week 104: Bodily pain | 1.6 (11.2) | 0.1 (8.5)
  Week 26: General health: number analyzed (Participants) | 482 | 465
  Week 26: General health | 2.5 (8.2) | 2.1 (7.6)
  Week 104: General health: number analyzed (Participants) | 335 | 190
  Week 104: General health | 2.3 (8.7) | 2.1 (8.3)
  Week 26: Vitality: number analyzed (Participants) | 482 | 465
  Week 26: Vitality | 1.4 (8.1) | 1.4 (8.0)
  Week 104: Vitality: number analyzed (Participants) | 335 | 190
  Week 104: Vitality | 1.5 (8.4) | 1.5 (8.0)
  Week 26: Social functioning: number analyzed (Participants) | 482 | 465
  Week 26: Social functioning | 1.8 (8.1) | 0.9 (8.8)
  Week 104: Social functioning: number analyzed (Participants) | 335 | 190
  Week 104: Social functioning | 0.9 (8.9) | 1.1 (7.6)
  Week 26: Role-emotional: number analyzed (Participants) | 482 | 465
  Week 26: Role-emotional | 0.6 (8.9) | 0.7 (8.8)
  Week 104: Role-emotional: number analyzed (Participants) | 335 | 190
  Week 104: Role-emotional | 1.6 (10.1) | 1.2 (8.2)
  Week 26: Mental health: number analyzed (Participants) | 482 | 465
  Week 26: Mental health | 1.7 (8.7) | 1.3 (8.4)
  Week 104: Mental health: number analyzed (Participants) | 335 | 190
  Week 104: Mental health | 2.5 (9.4) | 0.3 (8.9)
  Week 26: PCS: number analyzed (Participants) | 482 | 465
  Week 26: PCS | 1.6 (6.3) | 0.9 (6.3)
  Week 104: PCS: number analyzed (Participants) | 335 | 190
  Week 104: PCS | 1.0 (7.2) | 0.8 (6.0)
  Week 26: MCS: number analyzed (Participants) | 482 | 465
  Week 26: MCS | 1.3 (8.2) | 1.2 (8.0)
  Week 104: MCS: number analyzed (Participants) | 335 | 190
  Week 104: MCS | 2.0 (9.0) | 1.0 (7.8)

54. Secondary Outcome: Change in TRIM-D
Description: Treatment related impact measures-diabetes (TRIM-D) was developed according to the FDA guidance from 2009 on development of new PRO measures. The questionnaire consists of 5 sub-domains, which are scored according to a 1-5 point scale with a higher score indicating a better health state (less negative impact). Sub-domain scores are calculated by summing across items in the same sub-domain, and the total score is calculated by summing scores from all the sub-domains. The highest possible summed score within a sub-domain ranges from 20 (compliance sub-domain) to 40 (psychological health sub-domain) points and the highest possible total score is 140 points. Change in TRIM-D total score from baseline (week 0) to week 26 and week 104 is presented. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 26, week 104
Population: FAS included all randomised participants. 'Number analyzed'=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
Number analyzed (Participants) | 506 | 506
Score on a scale
  Week 26: number analyzed (Participants) | 477 | 456
  Week 26 | 9.6 (12.4) | 7.3 (13.1)
  Week 104: number analyzed (Participants) | 332 | 183
  Week 104 | 11.4 (13.7) | 9.5 (12.8)

ADVERSE EVENTS:
Time Frame: Weeks 0-104 (treatment period) + 7 days follow-up-1 + 30 days follow-up-2
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product administration. Results are based on the SAS which included all participants receiving at least one dose of trial product.
Arm/Group | Insulin Degludec/Liraglutide | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 2/506 | 5/504
Serious Adverse Events (participants affected / at risk) | 60/506 | 43/504
Other Adverse Events (participants affected / at risk) | 206/506 | 156/504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=506) | Insulin Glargine (N=504)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Angina unstable (Cardiac disorders) | 4 (4) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 0 (0)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tympanoplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=506) | Insulin Glargine (N=504)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (27) | 29 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (30) | 27 (40)
Diarrhoea (Gastrointestinal disorders) | 39 (52) | 12 (14)
Headache (Nervous system disorders) | 58 (98) | 45 (89)
Influenza (Infections and infestations) | 36 (46) | 28 (38)
Nasopharyngitis (Infections and infestations) | 57 (71) | 44 (53)
Nausea (Gastrointestinal disorders) | 31 (39) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 28 (30) | 36 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02501161/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02501161/SAP_001.pdf